CLINICAL TRIAL: NCT00568763
Title: Endogenous Heat-shock Vaccines for Melanoma A Feasibility Study
Brief Title: Radiofrequency Therapy-Induced Endogenous Heat-Shock Proteins With or Without Radiofrequency Ablation or Cryotherapy in Treating Patients With Stage IV Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000579004; P30CA015083 (NIH); MC0474 (Other: Mayo Clinic Cancer Center); 1189-05 (Other: Mayo Clinic IRB); NCI-2009-01304 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-12-05; First posted 2007-12-06 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — sargramostim; Immunoenzyme Techniques; Immunohistochemistry; Immunologic Techniques; Biopsy; Cryosurgery; Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: sargramostim
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: immunologic technique
Other: laboratory biomarker analysis
Procedure: biopsy
Procedure: cryosurgery
Procedure: radiofrequency ablation

SUMMARY:
RATIONALE: Radiofrequency therapy and radiofrequency ablation use a high-frequency electric current to kill tumor cells. Radiofrequency therapy can also cause the body to produce heat-shock proteins which may help kill more tumor cells. Cryotherapy kills tumor cells by freezing them. It is not yet known whether heat-shock proteins caused by radiofrequency therapy given together with radiofrequency ablation or cryotherapy is more effective in treating stage IV melanoma than radiofrequency therapy-induced heat-shock proteins alone.

PURPOSE: This randomized clinical trial is studying the side effects of radiofrequency therapy-induced endogenous heat-shock proteins when given alone or together with radiofrequency ablation or cryotherapy in treating patients with stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of endogenous heat-shock protein (hsp)70 synthesis at the site of the tumor using radiofrequency therapy (RFT) in patients with stage IV malignant melanoma.
* Determine the safety and feasibility of hsp70 release into the circulation using RFT alone vs RFT followed by radiofrequency ablation (RFA) or cryotherapy in these patients.
* Determine the feasibility of inducing a primary antitumor immune response using RFT with or without additional local therapy (i.e., RFA or cryotherapy) in these patients.
* Gain preliminary insight into the antitumor efficacy of an in vivo heat shock vaccine in these patients.

OUTLINE: Patients are randomized to 1 of 3 arms.

* Arm I (closed to enrollment as of 12/7/06): Patients undergo percutaneous biopsy of the target lesion and placement of a localization marker. Patients then undergo radiofrequency therapy (RFT) to the target lesion to induce the production of endogenous heat-shock proteins. After the procedure is completed, patients undergo a second biopsy of the target lesion. Patients also receive an intratumoral injection of sargramostim (GM-CSF) to promote further ablation at the tumor site.
* Arm II: Patients undergo percutaneous biopsies and RFT as in arm I followed by radiofrequency ablation of the target lesion. Patients also receive intratumoral GM-CSF as in arm I.
* Arm III: Patients undergo percutaneous biopsies and RFT as in arm I followed by cryoablation of the target lesion. Patients also receive intratumoral GM-CSF as in arm I.

Tumor tissue samples are obtained by core biopsy immediately before and immediately after RFT for RNA and protein analysis. Tissue samples are assessed by immunohistochemistry for tumor phenotype (i.e., MART-1, tyrosinase, or gp100) and for quantification of infiltrating lymphocytes. Peripheral blood samples are also obtained before and after treatment and periodically during study for immunologic analyses. Peripheral blood-derived lymphocytes are tested with a panel of monoclonal antibodies to estimate the percentages of cytotoxic T lymphocytes (CTLs), including CD4+ and CD8+ T cells as well as B cells, monocytes, and dendritic cells. In addition, assays are performed to estimate T-cell responses to polyclonal stimulus (i.e., PHA), recall antigens (i.e., tetanus toxoid), and HLA alloantigens. Estimates of peptide-specific CTLs are also obtained by enzyme-linked immunosorbent spot assays after in vitro stimulation with peptide-sensitized stimulator cells. Antibodies to extractable nuclear antigens (ENA) and antinuclear antibodies (ANA) will also be evaluated. GM-CSF levels and Hsp70 is assessed in tumor cells and peripheral blood by flow cytometry or enzyme-linked immunosorbent assays.

After completion of study therapy, patients are followed periodically for up to 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma meeting the following criteria:

  * Stage IV disease
  * Needle/probe accessible lesions of metastatic melanoma evident in the liver (or soft tissue) measuring 2 to 5 cm in size
  * HLA-A2 positive
* No known standard therapy that is potentially curative or proven capable of extending life expectancy

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 12 weeks
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Hemoglobin ≥ 10.0 g/dL
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine ≤ 1.5 times ULN
* Prothrombin time ≤ ULN
* Activated partial thromboplastin time ≤ ULN
* No uncontrolled or current infection
* No symptomatic heart disease (i.e., New York Heart Association classification III or IV)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No known immune deficiency

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior chemotherapy and recovered
* More than 4 weeks since prior immunotherapy, biologic therapy, or radiotherapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2005-11-25 (Actual); Primary Completion 2010-05-10 (Actual); Study Completion 2018-05-24 (Actual)

PRIMARY OUTCOMES:
Toxicity
Heat-shock protein levels
Tumor-specific immune response
Extent of lymphocyte infiltration
Tumor response by RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir N Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic Cancer Center, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Domingo-Musibay E, Heun JM, Nevala WK, Callstrom M, Atwell T, Galanis E, Erickson LA, Markovic SN. Endogenous Heat-Shock Protein Induction with or Without Radiofrequency Ablation or Cryoablation in Patients with Stage IV Melanoma. Oncologist. 2017 Sep;22(9):1026-e93. doi: 10.1634/theoncologist.2017-0060. Epub 2017 Jul 5. PMID 28679643